CLINICAL TRIAL: NCT05722587
Title: Students' Understanding and Beliefs About Pain Before and After a One-day Pain Science Education Conference: a Mixed-methods Evaluation
Brief Title: Students' Understanding and Beliefs About Pain Before and After a One-day Pain Science Education Conference: an Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Mrs Jagjit Mankelow, Lecturer in Rehabilitation Science, Teesside University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022 Oct 11360 Mankelow
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Pain, Chronic
Keywords: pain knowledge; pain beliefs; pain behaviour; experience of intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: multi site, non-randomised controlled, mixed methods study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain education day (Experimental): Pain education day, lecture and experiential
  Interventions: Other: Pain science education
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Pain science education — High school students receiving a day of pain science education in multiple formats, lectures, experiential, completing a task which consolidates the information.
  Other Names: Pain neuroscience education
  Arms: Pain education day

SUMMARY:
The beliefs held by students lead to behaviours in response to their pain which can be both helpful or a hindrance to how they manage their pain. The one-day education event aims to educate the cohort on the contemporary scientific understanding of persistent pain using a mixture of methods. It is hoped this event will result in an improvement in the alignment of beliefs and behaviours to contemporary understanding of persistent pain.

The principal aim is to evaluate the pre-post knowledge and beliefs about pain following a one-day pain education event in year 12 students, aged 16 or above.

DETAILED DESCRIPTION:
The students will be asked to complete questionnaires three times relating to their understanding and beliefs relating and intended behaviour in the presence of pain. Once at the start of the conference and once at the end, then finally after 3 months. The questionnaire will gather demographic information (age, gender, ethnicity and any history of persistent pain). There will also be a series of multiple-choice questions relating to knowledge and beliefs about persistent pain. The three time points of questionnaire completion will see the students complete the same questionnaire except they will not have to repeat demographic questions. The questionnaire should take 5-10 minutes to complete each time. The questionnaires will be provided online and links will be provided to participants.

This is a non-randomised controlled trial and a second school selected as it is part of the same group of schools and equally matched according to the English Indices of Deprivation 2019. This school will complete the survey at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Students at two specified schools in North Yorkshire who had been offered the pain study day in year 12 or are in the intervention or control school in year 12 or 13
* Aged above 16.
* Providing consent to participate.

Exclusion Criteria:

* Students not providing consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire (PBQ) | 3 months
  Helps to identify if participant beliefs are biomedical or biopsychosocial focussed, 12-item (Edwards et al, 1992, Walsh and Radcliffe, 2002). There are 2 scales within the PBQ: the organic beliefs scale has 8 items, with score ranges from 8-48, lower scores indicate less biomedical views and higher scores indicate more biomedical views. The psychological scale within the PBQ has 4 items with a score range of 4-24, a higher score indicates more biopsychosocial beliefs about pain and a lower score indicates less biopsychosocial beliefs.

SECONDARY OUTCOMES:
Concept of Pain Inventory-Adult (COPI-Adult) | 3 months
  The Concept of Pain Inventory-Adult was designed for assessing knowledge and beliefs about pain science (Pate et al, 2022). It is a 13-item questionnaire. Higher COPI-Adult scores reflect greater alignment with contemporary pain science (Total scores can range from 0-52).

OTHER OUTCOMES:
Vignette | 3 months
  Participants will be asked what actions they would take if they had pain with regards to medication, scans, daily activity, exercise and work either based on yes/no answers or four to five multiple choice answers. The percentage of recommendations in keeping with guidelines were measured from 0-100% with lower scores indicating intended behaviours that were not in keeping with guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom